CLINICAL TRIAL: NCT03526484
Title: The Utility of Urinalysis Prior to In-Office Procedures: A Randomized Clinical Trial
Brief Title: The Utility of Urinalysis Prior to In-Office Procedures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2017-1124; Protocol Version 5/28/2020 (Other: UW Madison); A539998 (Other: UW Madison); SMPH\VOLUNTEER STAFF\UROLOGY (Other: UW Madison)
Record Dates: First submitted 2018-05-03; First posted 2018-05-16 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Urinary Tract Infections
Keywords: UTI; Urinalysis; Urine Culture; Cystoscopy; BCG treatment; Prostate Biopsy
MeSH Terms: conditions — Urinary Tract Infections | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care (Active Comparator): The control group will have a urine sample taken for a urinalysis prior to their procedure, which will have a reflex urine culture done if urinalysis results are positive. The results of the urinalysis will be reported to the doctor performing the procedure. The provider may require participants to take antibiotics and/or delay their procedure as a result of the urinalysis.
  Interventions: Behavioral: Standard of Care
- Experimental (Experimental): The experimental group will have a urine sample taken for a urinalysis prior to their procedure, which will have a reflex urine culture done if urinalysis results are positive. The results of the urinalysis will NOT be reported to the doctor performing the procedure. Instead, the provider will conduct the procedure without looking at or acting upon the results of the urinalysis. The urinalysis and urine culture results will be monitored by the research team, and the participant will be informed if the urine culture results are positive for an infection.
  Interventions: Behavioral: Experimental

INTERVENTIONS:
Behavioral: Standard of Care — The provider will review the urinalysis results prior to conducting the in-office procedure and will make clinical decisions taking into account those results.
  Arms: Standard of Care
Behavioral: Experimental — The provider will not review the urinalysis results prior to conducting the in-office procedure, and therefore will not make clinical decisions taking those results into account.
  Arms: Experimental

SUMMARY:
The primary focus of this randomized clinical trial is to assess the usefulness of urinalysis prior to in-office urology procedures.

DETAILED DESCRIPTION:
OVERVIEW:

Current urology practice requires every patient to have a urinalysis lab done prior to any in-office procedures. If the patient's urinalysis is positive, they are then required to have a urine culture done, which takes 1-3 days to show results, and they may also be prescribed antibiotics. This practice may cause diagnostic delays, unnecessary cancellations of procedures, and the overuse of antibiotics.

The aim of this study is to assess the usefulness of urinalysis labs and urine cultures in patients prior to in-office cystoscopies, intravesical BCG treatments, and prostate biopsies. The investigators predict there is no difference in the number of cases of urinary tract infections in patients that undergo in-office procedures with or without a prior urinalysis. The investigators propose a change in protocol could allow for improved clinical efficiency, antibiotic stewardship, and be economically advantageous.

OUTLINE:

Participants will be randomly assigned to either receive standard of care before their procedure or have their procedure conducted by their provider without consulting the urinalysis results beforehand. Participants will have follow up questionnaires seven days and thirty days after their procedure. A total of 664 participants will be enrolled between the two study sites.

ELIGIBILITY:
Inclusion Criteria:

• Patients receiving an in office cystoscopy, intravesical BCG treatment, or prostate biopsy

Exclusion Criteria:

* Patients under 18
* Patients with symptomatic UTI infections at the time of recruitment
* Patients on antibiotics at the time of recruitment, not including prophylaxis
* Patients with a history of UTI within 1 year
* Patients with indwelling catheters
* Patients with clean intermittent catheterization
* Patients undergoing stent removals or with ureteral stents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2018-09-28 (Actual); Primary Completion 2021-11-15 (Actual); Study Completion 2021-11-15 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients who Developed a Urinary Tract Infection Post Procedure | 1 year
  Will compare difference in overall UTI rate between control and experimental groups.The results of the trial will be analyzed using a T-test for comparison of means, a Mann-Whitney U test for comparison of medians, Fisher's exact and chi-squared tests for comparison of categorical variables, and a logistic regression for predictors of UTI.

CONTACTS AND LOCATIONS:
Overall Officials: Kyle A Richards, MD, Principal Investigator — University of Wisconsin, Madison
Locations (2):
- United States (2):
  - William S. Middleton Memorial Veterans Hospital, Madison, Wisconsin
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-09-24): https://cdn.clinicaltrials.gov/large-docs/84/NCT03526484/Prot_SAP_001.pdf
  • Informed Consent Form (2018-06-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03526484/ICF_000.pdf